CLINICAL TRIAL: NCT06836661
Title: Effect, Cost, and sustaiNability of a Synergistic, Multipronged, Customized, Low-cost Intervention Package to Reduce cArdiovascular Burden Across India: a cLustEr RCT
Brief Title: Impact, Cost, and Sustainability of a Customized, Low-Cost Intervention to Reduce Cardiovascular Disease Burden in India: A Cluster Randomized Trial
Acronym: ENABLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Assam Medical College, Dibrugarh, India (Unknown); SRM Medical College Hospital & Research Centre (Unknown); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); Indian Council of Medical Research (Other Government); All India Institute of Medical Sciences, Bhopal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 293/2023
Record Dates: First submitted 2025-02-01; First posted 2025-02-20 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-02

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction of Anterior Wall; Cardiovascular Diseases
Keywords: CVD; Low cost intervention; task sharing; fixed dose combination pills
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Level 1: Patient
  1. Rational FDCs
  2. NPHWs and PMs mediated therapeutic lifestyle changes
  3. Texts/ WhatsApp reminders Level 2: Physician
  1. Reinforcing task sharing 2. Providing evidence on FDCs 3. Theory based behavior modification Level 3: Health administrators
  1. Pharmacy - Update drug formulary FDCs
  2. CV health days
  3. Facility strengthening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm - FDC and TLC and medication adherance (Experimental): NPHW enabled education and counseliing along with prescribing combination therapies and TLC and availability of low cost rational FDC at hospital pharmacy
  Interventions: Behavioral: FDC and TLC and medication adherance
- Control arm - Patients will Enhanced Usual Care (EUC) (Experimental): Enhanced Usual Care (EUC) with periodic follow ups.
  Interventions: Behavioral: Patients will Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: FDC and TLC and medication adherance — Level 1: Patient 1. Rational FDCs 2. NPHWs and PMs mediated therapeutic lifestyle changes 3. Texts/ WhatsApp reminders Level 2:Physician 1. Reinforcing task sharing 2. Providing evidence on FDCs 3. Theory based behavior modification Level 3: Health administrators 1. Pharmacy - Update drug formulary FDCs 2. CV health days 3. Facility strengthening
  Arms: Intervention arm - FDC and TLC and medication adherance
Behavioral: Patients will Enhanced Usual Care (EUC) — Patients will Enhanced Usual Care (EUC) with periodic follow ups
  Arms: Control arm - Patients will Enhanced Usual Care (EUC)

SUMMARY:
The ICRAG-2 project aims to assess the impact, cost-effectiveness, and sustainability of a low-cost, multipronged intervention package to reduce cardiovascular disease (CVD) burden in India. Given the high CVD mortality rate in India, this study addresses the urgent need for scalable, evidence-based solutions. The project will unfold in three steps: first, formative research including systematic reviews, cross-sectional studies, and qualitative studies will identify key barriers, facilitators, and refine interventions. Next, a matched-pair cluster randomized controlled trial (CRCT) across 26 clusters will evaluate the intervention's impact on CVD outcomes over three years, focusing on therapeutic lifestyle changes, fixed-dose medications, and task-sharing with non-physician health workers. Finally, the project will engage stakeholders through policy dialogues to support potential national-scale implementation. This trial offers a promising model to reduce CVD incidence through customized, sustainable interventions targeting patients, providers, and the health system.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the leading cause of death worldwide, responsible for approximately 17.9 million deaths each year, which accounts for 31% of all global deaths. The majority of these deaths-about 85%-are due to heart attacks and strokes. In India, CVD has contributed to 28·1% of the total deaths and 14·1% of the total DALYs. There is a remarkably high burden of CVD in India, with an age-standardised death rate of 282 deaths/100,000 (264-293) compared with global levels (233 deaths per 100,000 (229-236). Ischemic heart disease and stroke have been identified as the top two causes of mortality in the country, highlighting the urgent need for effective interventions.

Evidence supports the effectiveness of fixed dose combination treatments and the use of Non-Physician Health Workers (NPHWs) in primary and secondary prevention of CVD. India's healthcare system faces the dual challenge of rising CVD mortality and a lack of integrated preventive and management strategies for CVD at both the primary and secondary care levels. NPHWs play a major role in reducing CVD risk factors.

Despite the growing burden of CVD, there is a notable lack of evidence in India that evaluate comprehensive CVD management strategies across multiple levels, particularly focusing on hard clinical endpoints such as mortality, myocardial infarction (MI), stroke, and cardiovascular hospitalisations. To fill these gaps, we need a robust implementation trial that evaluates the effectiveness of multiple proven interventions in diverse settings on hard clinical endpoints. Such a trial, likely the first of its kind, would provide key evidence to guide policy decisions to improve CVD management strategies in India.

ELIGIBILITY:
Inclusion Criteria:

- 1. High-risk primary prevention A. Patients aged more than 40years of any gender without a CVD event (MI, Stroke) with at least two of the following risk factors, A to E with a 10 year documented evidence OF (a to d) a. Diabetes Mellitus b. Hypertension c. Dyslipidaemia d. Microalbuminuria e. Family history of premature CVD event (MI, stroke or CVD-related death under 55 years) B. Patients aged above 50years of any gender without a CVD event (MI, Stroke) with at least one year of documented disease, at least two A to D (Above) 2. High-risk secondary prevention Patients aged above 40 years or above, with a CVD event with any one of the following: options a. MI or stroke less than three months, <br/> b. MI or stroke, more than three months, but less than one year with at least one comorbid condition, that is A to E (Above).

c. Patients aged above 60 years or above with MI or stroke greater than three months BUT less than one year, without any comorbid condition. These patients are expected to have a moderate to high risk of a CVD event or death in the next three years.

Exclusion Criteria:

* We will exclude patients with any ONE of the following:

  1. Severe cognitive impairment of any aetiology and have no reliable caregivers.
  2. Medical conditions with a survival prognosis of less than 12 months.
  3. Unable to follow-up for the study period

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of death, myocardial infarction, stroke and CVD-related hospitalisations at three years | 3 years

SECONDARY OUTCOMES:
The Cost-Effectiveness (incremental cost- effectiveness ratio, ICER) of the IP | 3 years
  b) The Cost-Effectiveness (incremental cost- effectiveness ratio, ICER) of the IP c) Key Fidelity Metrics - utilisation rates of fixed-dose combinations, adherence to drug therapy at 12 months, proportion monitoring BP at home, adherence to different components of TLC and optimal referral.
  d) Key Implementation Metrics using the Reach Effectiveness-Adoption Implementation and Maintenance (RE-AIM) framework (Implementation research metric/ framework)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Xavier, Dr., Principal Investigator — St. John's Medical College and research Institute
Locations (1):
- Division of Clinical Research and training St. John's Research Institute Koramangala , - , India, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in specific publication arising out of the trial, after de-identiﬁcation (text, tables, ﬁgures, and appendices).